CLINICAL TRIAL: NCT04808180
Title: Effects of Biomimetic Hydroxyapatite in the Treatment of Molar Incisor Hypomineralization: a Randomized Clinical Trial.
Brief Title: Clinical Efficacy of Biomimetic Hydroxyapatite in the Treatment of Molar Incisor Hypomineralization.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-MIH
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Molar Incisor Hypomineralization
Keywords: biomimetic hydroxyapatite; enamel remineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Teeth from this group suffer from MIH. They will be evaluated after home oral care with BioRepair toothpaste containing microRepair®.
  Interventions: Other: Biorepair Shock Treatment
- Control Group (Active Comparator): Teeth from this group suffer from MIH. They are in the contralateral quadrants in respect to teeth from trial group. They will not be treated with the hydroxyapatite toothpaste.
  Interventions: Other: No treatment

INTERVENTIONS:
Other: Biorepair Shock Treatment — Teeth from this group will undergo the application of Biorepair Toothpaste for the first 7 days of the month for 9 months (1 application per day that lasts 10 minutes).
  Arms: Trial Group
Other: No treatment — Teeth from this group will not be treated with the experimental toothpaste.
  Arms: Control Group

SUMMARY:
The aim of the following study is to evaluate che clinical efficacy of a toothpaste with biomimetic hydroxyapatite for the management of Molar-Incisor Hypomineralization. Patients who agree to participate to the study will use Biorepair toothpaste for the first 7 days of the month for 3, 6 and 9 months. The following indices will be measured: BEWE, Bleeding Index, Gingival index, Plaque index and the dental sensitivity test. The contralateral tooth will be used as control if not affected by MIH; otherwise, adjacent teeth will be considered.

DETAILED DESCRIPTION:
Informed consent will be signed by the parents of the patients underage; patients will be asked the approval for the attendance of the study.

Adult patients will sign the informed consent for the treatment and for processing personal data for research purpose, with their approval for the attendance of the study.

Patients will be given for free a toothpaste with biomimetic hydroxyapatite (Biorepair Enamel-Repair Shock Treatment) and the Investigator will explain the correct procedures for home oral care. The toothpaste will be applied the first 7 days of the month for 9 months with a specific tray.

Teeth will be randomly assigned to:

* Trial group: 1 tooth with MIH from 1 quadrant will be treated with the biomimetic hydroxyapatite toothpaste. The applications will be performed for the first 7 days of the month for 9 months (1 application per day that lasts 10 minutes).
* Control group: 1 contralateral tooth with MIH will not be treated with the biomimetic hydroxyapatite toothpaste Patients will be visited after 1, 2, 3, 6 and 9 months from the baseline. For each visit, BEWE index, Bleeding Index, Gingival index, Plaque index and Dental sensitivity test. Tooth with MIH will be assessed, together with its contralaterals as control. If the contralateral tooth should suffer from MIH too, measurements will be carried out on the adjacent tooth.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least 2 enamel demineralizations of permanent molars and incisors (Molar-Incisor Hypomineralization - MIH) in contralateral quadrants
* good general health (absence of systemic diseases)

Exclusion Criteria:

* patients undergoing orthodontic therapy
* patients taking drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change of BI - Bleeding Index | Study begin, 1,2,3, 6 and 9 months
  Scoring criteria:
  * 0: absence of bleeding after 30 seconds
  * 1: bleeding observed after 30 seconds
  * 2: immediate bleeding
Change of GI - Gingival Index (Loe and Silness, 1963) | Study begin, 1,2,3, 6 and 9 months
  Scoring criteria:
  * 0 = normal gingiva.
  * 1 = mild inflammation, edema and swelling; no bleeding.
  * 2 = moderate inflammation with edema, swelling and bleeding on probing.
  * 3 = severe inflammation with marked edema, redness tissues, ulceration and spontaneous bleeding.
Change of PCR - Plaque Control Record (O'Leary, 1972) | Study begin, 1,2,3, 6 and 9 months
  4 surfaces scored (mesial, distal, vestibular, labial/palatal) per tooth by means of plaque relevator.
  The Index is calculated multiplying the total number of surfaces with plaque per 100.
Change in Schiff Air Index - Dental sensitivity test | Study begin, 1,2,3, 6 and 9 months
  Scoring criteria:
  0. the subject did not respond to air blasting;
  1. the subject responded to air blasting;
  2. the subject responded to air blasting and requested discontinuation;
  3. the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change of BEWE Index - Basic Erosive Wear Examination (Barlet et al., 2008) | Study begin, 1,2,3, 6 and 9 months
  Scoring criteria:
  * 0: no erosive tooth wear;
  * 1: initial loss of surface texture;
  * 2: distinct defect, hard tissue loss < 50% of the surface area;
  * 3: hard tissue loss ≥ 50% of the surface area.
  Additionally, risk level for clinical management will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator